CLINICAL TRIAL: NCT04422821
Title: Flash Glucose Monitoring in Gestational Diabetes Mellitus: Study Protocol for a Randomized Controlled Trial
Acronym: FLAMINGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, AGATA MAJEWSKA, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 931156
Record Dates: First submitted 2020-05-31; First posted 2020-06-09 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; flash glucose monitoring; glycemia
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FreeStyle Libre™ (Experimental): FreeStyle Libre™ will comprise 50 pregnant women between 24-28 weeks of gestation, diagnosed with gestational diabetes mellitus, who will receive subcutaneous sensor for glucose monitoring (FreeStyle Libre™; Abbott Diabetes Care, Alameda, CA) for 4 weeks.
  Interventions: Device: Flash Glucose Monitoring
- iXell® (Active Comparator): iXell® will comprise 50 pregnant women between 24-28 weeks of gestation, diagnosed with gestational diabetes mellitus, who will monitor glycemia through use of standard glucose meter (iXell®; Genexo sp; Warsaw, Poland) for 4 weeks.
  Interventions: Device: Self-Monitoring of Blood Glucose

INTERVENTIONS:
Device: Flash Glucose Monitoring — Flash Glucose Monitoring FreeStyle Libre™ (Abbott Diabetes Care, Alameda, CA) sensor placed subcutaneously that will be applied for 14 days, then removed and changed for the second sensor for the next 14 days.
  Other Names: FreeStyle Libre™ (Abbott Diabetes Care, Alameda, CA)
  Arms: FreeStyle Libre™
Device: Self-Monitoring of Blood Glucose — Self-Monitoring of Blood Glucose with a standard glucose meter (iXell®; Genexo sp; Warsaw, Poland) performed through a skin-puncturing 4 times a day for 28 days.
  Other Names: iXell®; Genexo sp; Warsaw, Poland
  Arms: iXell®

SUMMARY:
Gestational diabetes mellitus (GDM) is glucose intolerance diagnosed for the first time in pregnancy. According to literature GDM affects 3-10% of pregnant women and is a risk factor for multiple maternal and fetal complications. During pregnancy GDM significantly increases the risk of fetal macrosomia, shoulder dystocia, birth trauma and Cesarean section. Furthermore, the long-term complications of GDM include increased risk of development of diabetes mellitus type 2 in the mother, as well as increased risk of obesity, diabetes and metabolic syndrome occurrence in their children. It has been well-documented that the risk of above-mentioned complications increases with the level of maternal hyperglycemia.

Proper glycemia control is one of the key elements in the effective treatment of GDM. Until recently, glucose monitoring was solely performed using glucose meters, which required multiple fingerpricks. Nowadays, due to the glycemia monitoring systems development, such as flash glucose monitoring (FGM), glucose levels may be measured less invasively through subcutaneous sensor application. As shown in one of the studies, FGM due to the ease of use, was 3 times more often applied as a method of glycemia control than SMBG. As a result, patients from FGM group had significantly better blood glucose control.

The main purpose of our study is to evaluate the impact of new method of glycemia control (FGM) on the efficacy of treatment of GDM. By analyzing results of this study, such as mean glycemia levels, number of women requiring insulin therapy and maternal-fetal perinatal outcomes the investigators will provide a scientific basis for more common use of FGM in the population of pregnant women affected by GDM.

DETAILED DESCRIPTION:
This is a randomized controlled trial performed at the 1st Department of Obstetrics and Gynecology of Medical University of Warsaw. The study will recruit 100 women at 24-28 weeks of gestation . Women diagnosed with GDM, who will meet the inclusion criteria, will be individually randomized to Flash Glucose Monitoring (n=50) or Self-Monitoring of Blood Glucose (n=50) group.

The study group will obtain instruction for using Freestyle Libre app to measure and collect glycemia results using a mobile phone.

The control group will be informed about proper use of glucose meters.

All participants will be obliged to measure fasting and 1-h postprandial glucose concentrations in a daily manner, together with once per week midnight measurement.

All participants will obtain dietary recommendations for gestational diabetes mellitus and recommendations about daily physical activity in pregnancy.

In order to assess daily physical activity all participants will obtain a wristband allowing for footsteps measurement.

An evaluation of patient's dietary habits will be based on Eating Assessment Test prepared by the Polish National Institute of Public Health - National Institute of Hygiene.

Clinical and laboratory results of the mother and their newborns will be collected for analysis during the course of pregnancy.

After delivery, at the follow-up visit research staff will retrieve maternal and neonatal outcomes from patients medical history.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* singleton pregnancy between 24-28 weeks of gestation
* gestational diabetes mellitus diagnosis

Exclusion Criteria:

* multiple pregnancy
* fetal malformations
* pre-gestational diabetes mellitus
* chronic or pregnancy-induced hypertension
* chronic renal or hepatic disease, in-vitro fertilization
* delivery <37 weeks of gestation
* pre-mature rupture of membranes
* placenta previa
* stillbirth
* smoking in pregnancy
* intake of medications including: methyldopa, tetracyclin, acetylosalicylic acid, acetaminofen, ibuprofen, L-dopa, tolazamide, tolbutamide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Mean glycemia results (fasting and 1-h postprandial glucose concentrations) | 28 days after the recruitment visit
  Glycemia results analysis according to Polish Society of Obstetricians and Gynecologists (PSOG) recommendations for gestational diabetes mellitus.

SECONDARY OUTCOMES:
Number of patients requiring insulin therapy | 2, 4 and 8 weeks after the recruitment visit
  Number of patients in each group requiring insulin therapy will by analyzed at the second, third and fourth follow-up visit.
Long-term glycemic control using blood HbA1c serum concentration | 4 and 8 weeks after the recruitment visit
  Difference in HbA1c serum concentration in each group will by analyzed at the third and fourth follow-up visit.
Number of hypoglycemia episodes (glucose concentration <70 mg/dl) during one month analysis | 0-4 weeks after the recruitment visit
  Number of hypoglycemia episodes in each group will by analyzed at third visit, to check whether there is a difference between the groups.
Physical activity during one month analysis | 0-4 weeks after the recruitment visit
  Number of footsteps walk per day in each group will by analyzed at the third follow-up visit.
Compliance with diet recommendations | 2, 4 and 8 weeks after the recruitment visit
  Diet assessment in each group will be performed at the second, third and fourth follow-up visit to check compliance with diet recommendations.
Gestational weight gain | 2, 4 and 8 weeks after the recruitment visit
  Gestational weight gain in each group will by analyzed at the second, third and fourth follow-up visit.
Mode of delivery (rate of vaginal delivery/ Cesarean section) | 24-72 hours after the delivery
  Rate of vaginal delivery versus cesarean section in each group will by analyzed at the fifth follow-up visit.
Fetal birth-weight | 24-72 hours after the delivery
  Fetal birth-weight in each group will by analyzed at the fifth follow-up visit.
Neonatal glycemia | 24-72 hours after the delivery
  Neonatal glycemia in each group will by analyzed at the fifth follow-up visit, to check the rate of neonatal hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Wielgoś, MD PhD, Prof., Study Director — Medical University of Warsaw
Locations (1):
- 1st Department of Obstetrics and Gynecology, Medical University of Warsaw, Warsaw, Starynkiewicza Sq. 1/3, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The deidentified participant data will become available upon publishing the protocol and results of the study. Study protocol will be available immediately following publication.
Access Criteria: The data will be provided on reasonable request for anyone after methodologically sound proposal (contact details: amajewska2@wum.edu.pl).

REFERENCES:
- [Background] Scott EM, Bilous RW, Kautzky-Willer A. Accuracy, User Acceptability, and Safety Evaluation for the FreeStyle Libre Flash Glucose Monitoring System When Used by Pregnant Women with Diabetes. Diabetes Technol Ther. 2018 Mar;20(3):180-188. doi: 10.1089/dia.2017.0386. Epub 2018 Feb 22. PMID 29470094
- [Background] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581
- [Background] Mancini G, Berioli MG, Santi E, Rogari F, Toni G, Tascini G, Crispoldi R, Ceccarini G, Esposito S. Flash Glucose Monitoring: A Review of the Literature with a Special Focus on Type 1 Diabetes. Nutrients. 2018 Jul 29;10(8):992. doi: 10.3390/nu10080992. PMID 30060632
- [Background] Dunn TC, Xu Y, Hayter G, Ajjan RA. Real-world flash glucose monitoring patterns and associations between self-monitoring frequency and glycaemic measures: A European analysis of over 60 million glucose tests. Diabetes Res Clin Pract. 2018 Mar;137:37-46. doi: 10.1016/j.diabres.2017.12.015. Epub 2017 Dec 24. PMID 29278709
- [Derived] Majewska A, Stanirowski PJ, Tatur J, Wojda B, Radosz I, Wielgos M, Bomba-Opon DA. Flash glucose monitoring in gestational diabetes mellitus (FLAMINGO): a randomised controlled trial. Acta Diabetol. 2023 Sep;60(9):1171-1177. doi: 10.1007/s00592-023-02091-2. Epub 2023 May 10. PMID 37160787
- [Derived] Majewska A, Stanirowski P, Wielgos M, Bomba-Opon D. Flash glucose monitoring in gestational diabetes mellitus: study protocol for a randomised controlled trial. BMJ Open. 2021 Mar 2;11(3):e041486. doi: 10.1136/bmjopen-2020-041486. PMID 33653744